CLINICAL TRIAL: NCT02293486
Title: Study of Pomegranate Juice in the Modulation of Oxidative Stress Markers in Endurance-based Athletes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Vitalgrana Pomegranate SL (Unknown)
Responsible Party: Principal Investigator, Néstor Vicente-Salar, PhD, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GRA 01
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Oxidative Stress
Keywords: Antioxidants; Protein Carbonylation; Malondialdehyde; Punicaceae; Athletic Performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Arm that followed all the protocols with the exception of the pomegranate juice intake.
- Pomegranate Juice (Experimental): Arm that followed all the protocols and the pomegranate juice intake.
  Interventions: Dietary Supplement: Pomegranate juice
- Pomegranate Juice Dilution (Experimental): Arm that followed all the protocols and the pomegranate juice dilution (1:1) intake.
  Interventions: Dietary Supplement: Pomegranate juice

INTERVENTIONS:
Dietary Supplement: Pomegranate juice — Intake of 200 ml of pomegranate juice or pomegranate juice dilution during 21 days after exercise.
  Other Names: Zumo de Granada Vitalgrana
  Arms: Pomegranate Juice; Pomegranate Juice Dilution

SUMMARY:
The purpose of this study is to evaluate modifications of plasma protein carbonyls and malondialdehyde levels in endurance-based athletes after three weeks of pomegranate juice consumption.

ELIGIBILITY:
Inclusion Criteria:

* Perform specific endurance training sessions
* More than 1 hour per session and more than 3 sessions per week
* Have participated recently in a half marathon or similar event

Exclusion Criteria:

* Intake of antioxidant or anti-inflammatory supplementation
* Present a chronic disorder
* Non-smoker
* No-alcoholic beverage consumption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Protein carbonyls levels changes in plasma | day 0 and 22
  Protein carbonyl derivatives were determined using an adaptation of the colorimetric method published in Levine et al. (1994) based in the formation of a stable 2,4-dinitrophenyl (DNP) hydrazone product after the addition of 2,4-dinitrophenylhydrazine (DNPH) to tha plasma. Protein carbonyls were calculated as nmoles·mg-1 protein
Malondialdehyde levels changes in plasma | day 0 and 22
  Malondialdehyde was determined by high pressure liquid chromatography (HPLC) with fluorescence detection according to the method described by Laporta et al. (2007). Malondialdehyde levels were calculated as nmoles·g-1 protein

SECONDARY OUTCOMES:
Blood biochemical parameters changes in plasma | day 0 and 22
  Blood biochemical parameters is a composite outcome measure consisting in circulating plasma glucose (mg·dL-1), HDL-cholesterol (mg·dL-1), triglycerides (mg·dL-1), ferritin (ng·mL-1), lactate (mg·dL-1), sodium (mEq·L-1), potassium (mEq·L-1), creatine kinase (U·L-1), aspartate aminotransferase (U·L-1) and alanine aminotransferase (U·L-1) were analyzed through biochemistry methods.
C-reactive protein levels changes in plasma | day 0 and 22
  Determination by immunoassay of C-reactive protein (ng·mL-1) levels in plasma.
Soluble E-selectin levels changes in plasma | day 0 and 22
  Determination by immunoassay of soluble E-selectin (ng·mL-1) levels in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Roche, PhD, Study Director — University Miguel Hernández

REFERENCES:
- [Result] Aviram M, Dornfeld L, Rosenblat M, Volkova N, Kaplan M, Coleman R, Hayek T, Presser D, Fuhrman B. Pomegranate juice consumption reduces oxidative stress, atherogenic modifications to LDL, and platelet aggregation: studies in humans and in atherosclerotic apolipoprotein E-deficient mice. Am J Clin Nutr. 2000 May;71(5):1062-76. doi: 10.1093/ajcn/71.5.1062. PMID 10799367
- [Result] Trombold JR, Reinfeld AS, Casler JR, Coyle EF. The effect of pomegranate juice supplementation on strength and soreness after eccentric exercise. J Strength Cond Res. 2011 Jul;25(7):1782-8. doi: 10.1519/JSC.0b013e318220d992. PMID 21659887